CLINICAL TRIAL: NCT01578694
Title: Characterization of Proteoglycan Depletion in Femoroacetabular Impingement With T1ρ MRI
Brief Title: Characterization of Proteoglycan Depletion in Femoroacetabular Impingement With T1ρ Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2007231-01H
Record Dates: First submitted 2010-08-19; First posted 2012-04-17 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Femoroacetabular Impingement; Cartilage, Articular; Hip Joint; MRI
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Group (Other): The patient group has been diagnosed by the surgeon as having femoro-acetabular impingement (FAI) of the hip and will undergo a magnetic resonance imaging (MRI) test, more specifically, T1-rho to examine articular cartilage.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)
- Control healthy volunteers (Other): The control group has not been diagnosed with any hip problems, but will undergo a magnetic resonance imaging (MRI) test, more specifically, T1-rho to examine articular cartilage.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — T1 rho MRI is a modified pulse sequence from the standard T1 sequence used in the clinical MRI.

SUMMARY:
Magnetic resonance imaging (MRI) has proven to be one of the best ways to image articular cartilage. A tremendous amount of research has focused on cartilage imaging with an emphasis of early-osteoarthritis (OA) characterization. One of the techniques which has shown great promise is the imaging technique called T1ρ . The advantage of this pulse sequence is that it is sensitive to proteoglycans (PG), a major macromolecule degraded in OA. The study objective is to determine if T1ρ can acutely assess PG content in femoroacetabular impingement (FAI) which may allow physicians to differentiate between normal and early-OA cartilage states in FAI patients.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is one of the best ways to image articular cartilage. One of the techniques which has shown great promise is the imaging technique called T1ρ (T1-rho). T1ρ is a modified pulse sequence from the standard T1 sequence used in the clinical MRI. Because the initial phases of arthritis occur at the molecular level, the main advantage of the T1ρ pulse sequence is that it is sensitive to proteoglycan. Proteoglycan is a molecule that is important to cartilage structure, and is lost as osteoarthritis develops. If we can show that this non-invasive tool can accurately assess cartilage damage and levels of proteoglycan, the clinical applications are numerous. The results can potentially help determine optimal surgical techniques and timing of surgical intervention to halt or slow the progression of arthritis, and will assist in the study of the effects of FAI and the success of the surgery performed to correct FAI.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Patient has been diagnosed by the surgeon as having femoro-acetabular impingement (FAI) of the hip)
* Group 1: Must meet all the following criteria: A) History and Physical Exam 1) Intermittent pain worse with activity 2) Positive impingement test (pain with flexion, adduction, and internal rotation of affected hip) B) X-ray 1) No signs of OA on plain radiological films (i.e. no osteophytes, no loss of joint space) 2) Non-spherical femoral head
* Group 2: Patient has not been diagnosed by the surgeon as having any hip problems.

Exclusion Criteria:

* Previous Hip Surgeries (Pelvic Osteotomies)
* Previous Hip Trauma
* History of Pediatric Hip Pathology: Slipped Capital Femoral Epiphysis or Hip Dysplasia
* Over the age of 40 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assess articular cartilage using T1rho MRI | Pre-op (within 6 weeks prior to surgery)
  To provide a detailed quantitative assessment of the sensitivity of T1rho in the characterization of proteoglycan depletion in patients with or without femoroacetabular impingement.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — University of Ottawa / The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Rakhra KS, Lattanzio PJ, Cardenas-Blanco A, Cameron IG, Beaule PE. Can T1-rho MRI detect acetabular cartilage degeneration in femoroacetabular impingement?: a pilot study. J Bone Joint Surg Br. 2012 Sep;94(9):1187-92. doi: 10.1302/0301-620X.94B9.29981. PMID 22933489
- [Result] Anwander H, Rakhra KS, Melkus G, Beaule PE. T1rho Hip Cartilage Mapping in Assessing Patients With Cam Morphology: How Can We Optimize the Regions of Interest? Clin Orthop Relat Res. 2017 Apr;475(4):1066-1075. doi: 10.1007/s11999-016-5011-0. PMID 27506970
- [Result] McGuffin WS, Melkus G, Rakhra KS, Beaule PE. Is the contralateral hip at risk in patients with unilateral symptomatic cam femoroacetabular impingement? A quantitative T1rho MRI study. Osteoarthritis Cartilage. 2015 Aug;23(8):1337-42. doi: 10.1016/j.joca.2015.03.018. Epub 2015 Mar 25. PMID 25819578